CLINICAL TRIAL: NCT05788679
Title: A Phase II Multicenter Single-armed Study Using Subject-specific Minimal Residual Disease Markers to Adopt Treatment After Allogeneic Stem Cell Transplantation for Subjects With Myelodysplastic Syndrome
Brief Title: A Study Using Subject-specific MRD to Adopt Treatment After HSCT for Subjects With MDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Nordic MDS Group (Network)
Responsible Party: Principal Investigator, Magnus Tobiasson, Coordinating investigator, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMDSG14B, part 2
Record Dates: First submitted 2023-01-27; First posted 2023-03-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia With Myelodysplasia Related Disease and < 30% Blasts; Mixed Myelodysplastic/Myeloproliferative Disease
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention in MRD positive patients (Experimental): Azacitidine and / or Donor lymphocytes or tapering of immune suppression
  Interventions: Drug: Azacitidine; Other: Donor lymphocytes; Other: Tapering of immune suppression

INTERVENTIONS:
Drug: Azacitidine — Azacitidine
Other: Donor lymphocytes — Donor lymphocytes in patients without immune suppression
Other: Tapering of immune suppression — Tapering of immune suppression in patients who are on immune suppressive drugs

SUMMARY:
The goal of this interventional study is to evaluate if pre-emptive intervention using Azacitidine and / or donor lymphocytes or tapering of immune suppression in measurable residual disease (MRD) positive subjects can prevent clinical relapse. Participants will undergo MRD surveillance and be subjected to intervention in case of MRD positivity. Results will be compared with NMDSG14B, part one, in which MRD was analyzed in included patients without recieving intervention.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent

* Age ≥ 18 years
* Subjects eligible for SCT
* Subjects having the disease MDS, mixed myelodysplastic/myeloproliferative syndrome or AML with myelodysplasia related dysplasia and 20-29% marrow blasts
* All female subjects of childbearing potential have to have negative pregnancy test within 2 weeks prior to inclusion to the study

Exclusion Criteria:

* No traceable genetic aberration identified either in screening next generation sequencing panel or next generation sequencing panel performed at diagnosis
* Uncontrolled hypertension, heart, liver, kidney related or other uncontrolled medical or psychiatric disorders
* Mental inability, reluctance or language difficulties that results in difficulty understanding the meaning of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical event defined as relapse or death within 1 year from first MRD+ sample | Within 1 year from first MRD+ sample

SECONDARY OUTCOMES:
Number of MRD+ patients achieving MRD negativity | From MRD positivity until 2y after transplantation
Incidence and severity of graft-versus host disease | From transplantation until 2y after transplantation
Safety, adverse events reporting | After start of Azacitidine until 30 days after last azacitidine injection
Relapse-free survival | From transplantation until 2y after transplantation
Overall survival | From transplantation until 2y after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Tobiasson, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Department of Hematology, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No